CLINICAL TRIAL: NCT03020563
Title: Does Liposomal Bupivacaine Provide Improved Pain Management for ORIF of Midshaft Clavicle Fractures?
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no longer necessary
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1611M99381
Record Dates: First submitted 2017-01-05; First posted 2017-01-13 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Clavicle Fracture
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine (Active Comparator): Time release Bupivacaine
  Interventions: Drug: Liposomal Bupivacaine
- Bupivacaine (Placebo Comparator): Immediate Acting Bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Liposomal Bupivacaine — Liposomal Bupivacaine
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine — Bupivacaine
  Arms: Bupivacaine

SUMMARY:
To determine whether liposomal bupivacaine wound infiltration decreases pain scores and narcotic use when compared to bupivacaine alone after open reduction internal fixation of midshaft clavicle fractures.

ELIGIBILITY:
Inclusion Criteria:

* Mid-shaft Clavicle Fracture treated with ORIF

Exclusion Criteria:

* Unable to be contacted for 72 hours post surgery
* Other concurrent surgical procedures
* Chronic narcotic user

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Pain Scale Averages between the two treatments | 72 hours post surgery
  Scale is based on 1-10 with 1 being the lowest pain and 10 being the highest pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No